CLINICAL TRIAL: NCT01282346
Title: Clinical Evaluation of the SOLX Gold Shunt for the Reduction of Intraocular Pressure (IOP) in Refractory Glaucoma
Brief Title: SOLX Gold Shunt for Refractory Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOLX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLX84
Record Dates: First submitted 2011-01-05; First posted 2011-01-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Glaucoma; Glaucoma, Open Angle
Keywords: Glaucoma shunt; Ocular implant; Gold; Trabeculectomy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

ARMS (1):
- SOLX Gold Shunt (Experimental)
  Interventions: Device: SOLX Gold Shunt

INTERVENTIONS:
Device: SOLX Gold Shunt — Single use implant

SUMMARY:
To establish the clinical performance of the SOLX Gold Shunt for its ability to reduce intraocular pressure (IOP) in eyes with refractory glaucoma where medical and conventional surgical treatments have failed.

ELIGIBILITY:
Inclusion Criteria:

* primary open-angle glaucoma
* age 21 or over
* refractory glaucoma, with IOP ≥ 24 mmHg on medications and failed prior incisional glaucoma surgery
* detectable visual field defect (negative MD score)
* written informed consent
* available for up to 24 months follow-up

Exclusion Criteria:

* either eye with VA worse than count fingers
* angle closure glaucoma episode within past 12 months
* uveitic glaucoma, iridocorneal endothelial (ICE) syndrome, traumatic glaucoma, or neovascular glaucoma
* diagnosis of pigmentary glaucoma or pseudoexfoliative glaucoma
* other significant ocular disease, except cataract
* active ocular infection
* expected ocular surgery in next 12 months
* no suitable quadrant for implant
* systemic corticosteroid therapy > 5 mg/day prednisone
* intolerance to gonioscopy or other eye exams
* mental impairment interfering with consent or compliance
* pregnancy
* known sensitivity to anticipated medications used at surgery
* significant co-morbid disease
* concurrent enrollment in another drug or device study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes that achieve an IOP of > 5mmHg and ≤ 21 mmHg, irrespective of medication use | 1 year

SECONDARY OUTCOMES:
Average change in IOP | 1 & 2 years
Percentage change in IOP from baseline | 1 & 2 years
Average change in number of glaucoma medications | 1 & 2 years
Visual acuity changes | 1 & 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Shah, MD, Study Director — The Emmes Company, LLC
Locations (17):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Vold Vision, PLLC, Springdale, Arkansas
  - University of California, Irvine, Irvine, California
  - Yale University, New Haven, Connecticut
  - Illinois Eye Institute, Chicago, Illinois
  - Glaucoma Associates of New York, New York, New York
  - Ophthalmic Partners of Pennsylvania, Bala-Cynwyd, Pennsylvania
  - University Eye Surgeons, Maryville, Tennessee
  - Glaucoma Associates of Texas, Dallas, Texas
  - University of Virginia, Charlottsville, Virginia
  - Memmen, Ltd, Green Bay, Wisconsin
- University of Campinas, Campinas, Brazil
- Canada (3):
  - Clarity Eye Institute, Vaughan, Ontario
  - Institut de l'oeil des Laurentides, Boisbriand, Quebec
  - Bellevue Ophthalmology Clinic, Montreal, Quebec
- Medical Research Infrastructure Department and Health Services Fund by the Sheba Medical Center (R.A.), Tel Litwinsky, Israel
- Centro Medico Docente La Trinidad, Caracas, Venezuela